CLINICAL TRIAL: NCT03076138
Title: The Clinical Trial of the Safety and Efficacy of the Medical Device "Bone Substitute Based on Octacalcium Phosphate and Biologically Active Nucleic Acids for Bone Tissue Regeneration" (Nucleostim-VEGF)
Brief Title: Gene-activated Bone Substitute for Maxillofacial Bone Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Histograft Co., Ltd. (Industry)
Collaborators: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-Histograft-20-08-2016
Record Dates: First submitted 2017-03-05; First posted 2017-03-10 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Bone Cysts; Bone Atrophy; Bone Deformity; Bone Fracture; Bone Loss; Tooth Loss
Keywords: Gene-activated matrix; Bone substitute; Bone grafting; Dental implantation; gene therapy; plasmid DNA; VEGF gene; octacalcium phosphate
MeSH Terms: conditions — Bone Cysts; Fractures, Bone; Bone Diseases, Metabolic; Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Bone grafting with gene-activated matrix (OCP + plasmid DNA with VEGF gene)
  Interventions: Device: Gene-activated matrix (OCP + plasmid DNA with VEGF gene)

INTERVENTIONS:
Device: Gene-activated matrix (OCP + plasmid DNA with VEGF gene) — Bone grafting procedure with investigated medical device

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the gene-activated bone substitute consisting of octacalcium phosphate and plasmid DNA encoding vascular endothelial growth factor (VEGF) for maxillofacial bone regeneration. The patients with congenital and acquired maxillofacial bone defects and alveolar ridge atrophy will be enrolled.

DETAILED DESCRIPTION:
All participants of the study will receive standard treatment according to the medical care standards for diseases and pathological conditions characterized by maxillofacial bone defects and/or alveolar ridge atrophy. Bone grafting procedures as part of the surgical treatment will be performed with the use of investigated medical device. The safety and efficacy of the implanted gene-activated bone substitute will be evaluated by clinical examination, comprehensive laboratory tests, and computer tomography within 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* obtained voluntary informed consent for participation in the clinical study;
* congenital and acquired maxillofacial bone defects (sockets of extracted teeth, bone defects after injuries, surgeries, removal of benign neoplasms and pseudotumors, etc.) or alveolar ridge atrophy.

Exclusion Criteria:

* not able or unwilling to give voluntary informed consent for the study or follow requirements of the clinical study;
* decompensated chronic visceral diseases;
* clinically significant laboratory abnormalities;
* HIV, HBV and HCV antibodies in serum;
* alcohol consumption within 4 days prior the study;
* history of drug addiction;
* participation in other clinical trials (or administration of study products) within 3 months prior the study;
* conditions limiting study compliance (dementia, psycho-neurological diseases, drug addiction, alcoholism, etc.);
* pregnancy or lactation;
* malignancies including post-treatment period (surgical, chemotherapy, radiation therapy both alone and in different combinations) less than 5 years prior the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Bone tissue formation in the field of gene-activated bone substitute implantation | 6 months
  To determine the quantity of newly formed bone tissue the following morphometric parameters will be measured on CT scan using special tools ("ROI", region of interest, etc.):
  * average density (in HU);
  * size (length, width, height) and volume.
  All together both measurements allow to determine "bone tissue formation" as a value derived from the presence of newly formed bone tissue and its volume correspondence with the quantity of the material implanted.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | 6 months
  Evaluation of the Adverse Events and Serious Adverse Events frequency
Surgical failure rate | 6 months
  Evaluation of the events frequency when the surgery was not completed due to the reasons related with gene-activated bone substitute

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Y. Drobyshev, MD,PhD,Prof., Principal Investigator — A.I. Evdokimov Moscow State University of Medicine and Dentistry
Locations (1):
- A.I. Moscow State University of Medicine and Dentistry, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Detailed results of the study will be published in a specialized peer-reviewed scientific journal with an open access

REFERENCES:
- [Background] Deev RV, Drobyshev AY, Bozo IY, Isaev AA. Ordinary and Activated Bone Grafts: Applied Classification and the Main Features. Biomed Res Int. 2015;2015:365050. doi: 10.1155/2015/365050. Epub 2015 Nov 15. PMID 26649300
- [Background] Komlev VS, Barinov SM, Bozo II, Deev RV, Eremin II, Fedotov AY, Gurin AN, Khromova NV, Kopnin PB, Kuvshinova EA, Mamonov VE, Rybko VA, Sergeeva NS, Teterina AY, Zorin VL. Bioceramics composed of octacalcium phosphate demonstrate enhanced biological behavior. ACS Appl Mater Interfaces. 2014 Oct 8;6(19):16610-20. doi: 10.1021/am502583p. Epub 2014 Sep 16. PMID 25184694
- [Background] Komlev VS, Popov VK, Mironov AV, Fedotov AY, Teterina AY, Smirnov IV, Bozo IY, Rybko VA, Deev RV. 3D Printing of Octacalcium Phosphate Bone Substitutes. Front Bioeng Biotechnol. 2015 Jun 8;3:81. doi: 10.3389/fbioe.2015.00081. eCollection 2015. PMID 26106596
- [Background] Deev R, Plaksa I, Bozo I, Isaev A. Results of an International Postmarketing Surveillance Study of pl-VEGF165 Safety and Efficacy in 210 Patients with Peripheral Arterial Disease. Am J Cardiovasc Drugs. 2017 Jun;17(3):235-242. doi: 10.1007/s40256-016-0210-3. PMID 28050885
- [Background] Deev RV, Bozo IY, Mzhavanadze ND, Voronov DA, Gavrilenko AV, Chervyakov YV, Staroverov IN, Kalinin RE, Shvalb PG, Isaev AA. pCMV-vegf165 Intramuscular Gene Transfer is an Effective Method of Treatment for Patients With Chronic Lower Limb Ischemia. J Cardiovasc Pharmacol Ther. 2015 Sep;20(5):473-82. doi: 10.1177/1074248415574336. Epub 2015 Mar 13. PMID 25770117